CLINICAL TRIAL: NCT00744718
Title: Bevacizumab and Carboplatin for Patients With Platin Resistant Epithelial Ovarian Cancer. A Phase II Study.
Brief Title: Bevacizumab and Carboplatin for Patients With Ovarian Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vejle Hospital (Other)
Responsible Party: Sponsor
Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 2008-000878-20; S-20080033; 2612-3754
Record Dates: First submitted 2008-08-29; First posted 2008-09-01 (Estimated); Last update posted 2016-11-16 (Estimated); Status verified 2016-11

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Bevacizumab; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Bevacizumab — Bevacizumab 10 mg/kg every 3 weeks
Drug: Carboplatin — Carboplatin AUC 5 every 5 weeks

SUMMARY:
This is a phase II trial to investigate the effect of bevacizumab and carboplatin in patients with platin resistant ovarian cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically verified epithelial ovarian cancer, primary tubae- or primary peritoneal cancer (Stage I-IV)
2. Carboplatin resistant ovarian cancer previously treated with a maximum of three different cytostatic regimens (single substance or in combination).
3. Age ≥ 18 years.
4. Performance status 0-2.
5. Measurable disease according to CA125 GCIG criteria (Gynaecologic Cancer Intergroup) or RECIST (Response Evaluation Criteria in Solid Tumors) (See appendix I+II)
6. Adequate bonemarrow, liver and kidney function and coagulation parameters (within seven days of start of treatment).
7. ANC ≥ 1.5*109
8. Thrombocytes ≥ 100*10^9/L
9. Haemoglobin (Hb) ≥ 6 mmol/l
10. Se-bilirubin (BR) ≤ 1.5*ULN (Upper Limit of Normal)
11. Se-transaminase ≤ 2.5*ULN
12. Se-creatinin ≤ 1.5*ULN
13. Urin stix for protein <2+ (If stix shows protein ≥2+ urin must be measured 24 hours where the protein content must be under 1 g.)
14. INR ≤1.5
15. APTT ≤ 1.5*ULN
16. Signed informed consent form.

Exclusion Criteria:

1. Patients who have received other types of experimental treatment or participated in a clinical study less than 28 days prior to this study.
2. Pregnant or breastfeeding women. A negative pregnancy test is mandatory for fertile women.
3. Fertile women, who do not wish to use safe contraception (e.g., birth control pills, coil, gestagen deposit injection, subdermal implantation, hormonal vagina ring, and transdermal deposit band-aid).
4. Untreated bowel obstruction or massive gastrointestinal tumors verified by CT scan.
5. Other present or previous malignant disease apart from curatively treated non-melanoma skin cancer or other types of cancer with minimal risk of relapse.
6. CNS-metastases.
7. Underlying medical disease not adequately treated (diabetes, cardiovascular disease).
8. Uncontrolled hypertension (persistent BP > 150/100 despite antihypertensive treatment).
9. Surgery incl. open biopsy less than 4 weeks before expected first dose of Bevacizumab.
10. Patients with non-healing wounds or fractures.
11. Previous cerebrovascular attack (TVA), transient ischaemic attack (TIA) or subarachnoidal bleeding (SAH) within last six months.
12. Thromboembolic or haemorrhagic disease in the anamnesis.
13. Clinically significant cardiovascular disease including Myocardial infarction or unstable angina less than 6 months prior to treatment

    * New York heart Association NYHA class ≥ 2
    * Poorly controlled cardial arrythmia despite medical treatment
    * Peripheral vascular disease, grade 3 or above.
14. Present or previous chronical use of Aspirin (less than 10 days before start of treatment) Aspirin > 325 mg daily.
15. Present or recent use of full dose oral or parenteral anticoagulant or thrombolytic medicine.
16. Preexisting neuropathy, sensoric or motoric ≥ grade 2.
17. Decreased hearing.
18. Bleeding tumor.
19. Hypersensitivity to the active substance or one or more of the other substances contained in the protocol drugs.
20. Hypersensitivity to products from ovarian cells (CHO) from Chinese hamster or other recombinant or humanized antibodies.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2008-08; Primary Completion 2015-08 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Progression free survival | From date of first treatment until date of verified progression or death. 12 months of follow-up

SECONDARY OUTCOMES:
Overall survival | From date of first treatment until death. Up to 12 months
Response rate | Every 9 weeks until progression or death. Up to 12 months
Response duration | From date of first documented response until date of progression. Up to 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Anders Jakobsen, MD, DMSc, Study Chair — Department of Oncology, Vejle Hospital
Locations (1):
- Vejle Hospital, Vejle, Denmark

REFERENCES:
- [Derived] Gaitskell K, Rogozinska E, Platt S, Chen Y, Abd El Aziz M, Tattersall A, Morrison J. Angiogenesis inhibitors for the treatment of epithelial ovarian cancer. Cochrane Database Syst Rev. 2023 Apr 18;4(4):CD007930. doi: 10.1002/14651858.CD007930.pub3. PMID 37185961